CLINICAL TRIAL: NCT05372731
Title: Recruitment Maneuver After Bronchoalveolar Lavage in ARDS Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Director of Intensive Care Unit, Principal Investigator, Clinical Professor, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BAL20220420
Record Dates: First submitted 2022-04-20; First posted 2022-05-13 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RM after BAL (Experimental): patients underwent RM after BAL
  Interventions: Other: Recruitment Maneuver
- Non-RM after BAL (No Intervention): patients did not undergo RM after BAL

INTERVENTIONS:
Other: Recruitment Maneuver — RM after BAL
  Arms: RM after BAL

SUMMARY:
ARDS caused by pneumonia is one of the main reasons for ICU admission in critically ill patients, and also a common complication in patients admitted to ICU with invasive mechanical ventilation. Bronchoalveolar lavage (BAL) is the main diagnostic method for these patients, which often leads to alveolar collapse and exacerbates hypoxemia. In clinical practice, recruitment maneuver (RM) is often used immediately after BAL to prevent such a situation, but there is a lack of data on RM after BAL.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with invasive mechanical ventilation;
2. Patients who diagnosed with ARDS according to the Berlin definition
3. There are indications for bronchoalveolar lavage

Exclusion Criteria:

1. Patients with contraindications for EIT procedures;
2. Patients with contraindications for RM;
3. Previous chronic respiratory diseases (long-term home oxygen therapy for chronic respiratory diseases such as pulmonary fibrosis or COPD);
4. Pregnancy;
5. Refusal to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-30 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
the ratio of tidal volume in the BAL side and the other side | up to 24 hours
  distribution of tidal volume monitored by electrical impedance tomography from the BAL side to the other side

SECONDARY OUTCOMES:
partial pressure of arterial oxygen (Pao2) to the fraction of inspired oxygen (Fio2) ratio | up to 24 hours
  partial pressure of arterial oxygen (Pao2) to the fraction of inspired oxygen (Fio2) ratio
respiratory system compliance (the tidal volume to the driving pressure ratio) | up to 24 hours
  respiratory system compliance was calculated by dividing expiratory tidal volume by the driving pressure (plateau pressure minus positive end-expiratory pressure)

CONTACTS AND LOCATIONS:
Overall Officials: ling liu, phD, Principal Investigator — Zhongda Hospital

IPD SHARING:
Plan to Share IPD: No